CLINICAL TRIAL: NCT06364410
Title: Phase 1 Study of Trastuzumab Deruxtecan (DS-8201a) in Combination With Azenosertib (ZN-c3) in HER2-Expressing/Amplified Cyclin E-Amplified Gastric/Gastroesophageal Junction Cancer and Other Solid Tumors With HER2 Expression
Brief Title: Testing the Combination of the Anticancer Drugs Trastuzumab Deruxtecan (DS-8201a) and Azenosertib (ZN-c3) in Patients With Stomach or Other Solid Tumors
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Other - Pending amendment.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2024-02982; NCI-2024-02982 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10554 (Other: University of Texas MD Anderson Cancer Center LAO); 10554 (Other: CTEP); UM1CA186688 (NIH)
Record Dates: First submitted 2024-04-12; First posted 2024-04-15 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Clinical Stage III Gastric Cancer AJCC v8; Clinical Stage III Gastroesophageal Junction Adenocarcinoma AJCC v8; Clinical Stage IV Gastric Cancer AJCC v8; Clinical Stage IV Gastroesophageal Junction Adenocarcinoma AJCC v8; Locally Advanced Gastric Carcinoma; Locally Advanced Gastroesophageal Junction Adenocarcinoma; Locally Advanced Malignant Solid Neoplasm; Metastatic Gastric Carcinoma; Metastatic Gastroesophageal Junction Adenocarcinoma; Metastatic Malignant Solid Neoplasm; Unresectable Gastric Carcinoma; Unresectable Gastroesophageal Junction Adenocarcinoma; Unresectable Malignant Solid Neoplasm
MeSH Terms: conditions — Stomach Neoplasms; Neoplasm Metastasis | interventions — Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; trastuzumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose escalation (T-DXd, azenosertib) (Experimental): Patients receive T-DXd IV over 30-90 minutes on day 1 of each cycle and azenosertib PO QD on days 1-5, 8-12, and 15-19 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo ECHO or MUGA and collection of blood samples at screening and on study and undergo CT or MRI throughout the trial.
  Interventions: Drug: Azenosertib; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Biological: Trastuzumab Deruxtecan
- Dose expansion, Cohort 1 (T-DXd, azenosertib) (Experimental): Patients receive T-DXd IV over 30-90 minutes on day 1 of each cycle and azenosertib PO QD on days 8-12 and 15-19 of cycle 1 and days 1-5, 8-12, and 15-19 in subsequent cycles. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo ECHO or MUGA and collection of blood samples at screening and on study and undergo CT or MRI throughout the trial. Patients also undergo biopsy at screening and on study.
  Interventions: Drug: Azenosertib; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Biological: Trastuzumab Deruxtecan
- Dose expansion, Cohort 2 (T-DXd, azenosertib) (Experimental): Patients receive treatment as in the dose escalation arm. Patients also undergo ECHO or MUGA and collection of blood samples at screening and on study and undergo CT or MRI throughout the trial. Patients also undergo biopsy at screening and on study.
  Interventions: Drug: Azenosertib; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Biological: Trastuzumab Deruxtecan

INTERVENTIONS:
Drug: Azenosertib — Given PO
  Other Names: Wee1 Inhibitor ZN-c3; ZN c3; ZN-c3; ZNc3
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
  Arms: Dose expansion, Cohort 1 (T-DXd, azenosertib)
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Biological: Trastuzumab Deruxtecan — Given IV
  Other Names: DS-8201; DS-8201a; Enhertu; Fam-trastuzumab Deruxtecan-nxki; T-DXd; WHO 10516

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of azenosertib in combination with trastuzumab deruxtecan in treating patients with HER2-positive and cyclin E amplified gastric or gastroesophageal junction cancer and other HER2-positive solid tumors that have spread to nearby tissue or lymph nodes (locally advanced), that have spread from where it first started (primary site) to other places in the body (metastatic), or that cannot be removed by surgery (unresectable). Azenosertib is in a class of medications called kinase inhibitors. It inhibits a protein called Wee1. Inhibition of the Wee1 protein can make tumor cells more vulnerable to chemotherapy drugs, leading to tumor cell death. Trastuzumab deruxtecan is in a class of medications called antibody-drug conjugates. It is composed of a monoclonal antibody, called trastuzumab, linked to a chemotherapy drug, called deruxtecan. Trastuzumab attaches to HER2 positive cancer cells in a targeted way and delivers deruxtecan to kill them. Giving azenosertib in combination with trastuzumab deruxtecan may be safe, tolerable, and/or more effective in treating patients with locally advanced, metastatic, or unresectable HER2-positive gastric, gastroesophageal junction, or other solid tumors, compared to just trastuzumab deruxtecan alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety and tolerability of trastuzumab deruxtecan (T-DXd; DS-8201a) in combination with azenosertib (ZN-c3) in human epidermal growth factor receptor 2 (HER2)-expressing/amplified solid tumors.

SECONDARY OBJECTIVES:

I. To observe and record the antitumor activity of the T-DXd (DS-8201a) and azenosertib (ZN-c3) combination.

II. To assess the pharmacodynamic effects of T-DXd (DS-8201a) in combination with azenosertib (ZN-c3).

III. To assess predictors of response and acquired resistance to the T-DXd (DS-8201a) and azenosertib (ZN-c3) combination.

OUTLINE: This is a dose-escalation study of azenosertib followed by a dose-expansion study.

DOSE ESCALATION: Patients receive T-DXd intravenously (IV) over 30-90 minutes on day 1 of each cycle and azenosertib orally (PO) once daily (QD) on days 1-5, 8-12, and 15-19 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo echocardiography (ECHO) or multigated acquisition scan (MUGA) and collection of blood samples at screening and on study and undergo computed tomography (CT) or magnetic resonance imaging (MRI) throughout the trial.

DOSE EXPANSION: Patients are assigned to 1 of 2 cohorts.

COHORT 1: Patients receive T-DXd IV over 30-90 minutes on day 1 of each cycle and azenosertib PO QD on days 8-12 and 15-19 of cycle 1 and days 1-5, 8-12, and 15-19 in subsequent cycles. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo ECHO or MUGA and collection of blood samples at screening and on study and undergo CT or MRI throughout the trial. Patients also undergo biopsy at screening and on study.

COHORT 2: Patients receive treatment as in the dose escalation arm. Patients also undergo ECHO or MUGA and collection of blood samples at screening and on study and undergo CT or MRI throughout the trial. Patients also undergo biopsy at screening and on study.

After completion of study treatment, patients are followed up at 30 days and then every 3 months in years 1 and 2 and every 6 months in year 3.

ELIGIBILITY:
Inclusion Criteria:

* In the dose escalation, patients must have a histologically documented locally advanced, unresectable, or metastatic solid tumor that has progressed following at least one prior line of treatment in the metastatic setting or has no satisfactory alternative treatment option and all of the following:

  * HER2 expression by immunohistochemistry (IHC) (1+, 2+, or 3+) or HER2 amplification by in situ hybridization (ISH) or next generation sequencing (NGS) (on any Clinical Laboratory Improvements Amendments [CLIA] platform), AND
  * T-DXd (DS-8201a)-naive disease
* In the dose expansion, patients must have histologically documented locally advanced, unresectable or metastatic gastric or gastroesophageal junction (GEJ) cancer that has progressed following at least one prior line of treatment in the metastatic setting and have all of the following:

  * CCNE1 amplification, AND
  * HER2 expression by IHC (1+, 2+, or 3+) or HER2 amplification by ISH or NGS (on any CLIA platform), AND
  * T-DXd (DS-8201a)-naive disease
  * Received prior trastuzumab-based treatment, if eligible for such treatment
* For the dose escalation and dose expansion, patients can have evaluable or measurable disease
* Potential trial participants should have recovered from clinically significant adverse events (AEs) of their most recent therapy/intervention prior to enrollment
* Age ≥ 18 years. Because no dosing or AE data are currently available on the use of T-DXd (DS-8201a) in combination with azenosertib (ZN-c3) in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1 (Karnofsky ≥ 70%). Both T-DXd (DS-8201a) and azenosertib (ZN-c3) have fatigue as an adverse effect. Due to the overlapping adverse effect, the performance status cannot be less restrictive
* Absolute neutrophil count ≥ 1.5 × 10^9/L (within 7 days of study treatment initiation)

  * No transfusions with red blood cells or platelets are allowed within 1 week prior to screening assessment
  * No administration of granulocyte colony-stimulating factor is allowed within 1 week prior to screening assessment
* Hemoglobin > 9.0 g/dL (within 7 days of study treatment initiation)

  * No transfusions with red blood cells or platelets are allowed within 1 week prior to screening assessment
  * No administration of granulocyte colony-stimulating factor is allowed within 1 week prior to screening assessment
* Platelets ≥ 100 × 10^9/L (within 7 days of study treatment initiation)

  * No transfusions with red blood cells or platelets are allowed within 1 week prior to screening assessment
  * No administration of granulocyte colony-stimulating factor is allowed within 1 week prior to screening assessment
* Total bilirubin ≤ 1.5 institutional upper limit of normal (ULN). Documented Gilbert syndrome is allowed if total bilirubin is ≤ 3 × institutional ULN (within 7 days of study treatment initiation)

  * No transfusions with red blood cells or platelets are allowed within 1 week prior to screening assessment
  * No administration of granulocyte colony-stimulating factor is allowed within 1 week prior to screening assessment
* Aspartate aminotransferase (AST [serum glutamic-oxaloacetic transaminase (SGOT)])/alanine aminotransferase (ALT [serum glutamate pyruvate transaminase (SGPT)]) ≤ 3 × institutional ULN. In the presence of liver metastases, AST or ALT up to 5 × institutional ULN is permitted (within 7 days of study treatment initiation)

  * No transfusions with red blood cells or platelets are allowed within 1 week prior to screening assessment
  * No administration of granulocyte colony-stimulating factor is allowed within 1 week prior to screening assessment
* Measured of calculated creatinine clearance (CrCl) ≥ 60 mL/min (CrCl should be calculated per institutional standard; glomerular filtration rate can also be used in place of CrCl) ≥ 60 mL/min for patients with creatinine levels > 1.5 x institutional ULN (within 7 days of study treatment initiation)

  * No transfusions with red blood cells or platelets are allowed within 1 week prior to screening assessment
  * No administration of granulocyte colony-stimulating factor is allowed within 1 week prior to screening assessment
* International normalized ratio/prothrombin time and activated partial thromboplastin time ≤ 1.5 × institutional ULN (within 7 days of study treatment initiation)

  * No transfusions with red blood cells or platelets are allowed within 1 week prior to screening assessment
  * No administration of granulocyte colony-stimulating factor is allowed within 1 week prior to screening assessment
* Patients must have left ventricular ejection fraction (LVEF) ≥ 50% by either an echocardiogram (ECHO) or multigated acquisition (MUGA) scan within 28 days before enrollment
* Human immunodeficiency virus-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression
* Patients with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate CNS-specific treatment is not required and is unlikely to be required during the first cycle of study treatment
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Life expectancy ≥ 3 months
* Women of childbearing potential (WOCBP) must have a negative serum pregnancy test result within 3 days of study treatment initiation
* Agents composed of HER2 antibody conjugated to a topoisomerase 1 inhibitor and azenosertib (ZN-c3) are known to be teratogenic; thus, WOCBP must agree to use highly effective contraception from time of screening and throughout the study treatment period and for at least 7 months after final study treatment administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Female patients must not donate, or retrieve for their own use, ova from the time of screening and throughout the study treatment period and for at least 7 months after the final study treatment administration
* Women of non-childbearing potential defined as premenopausal females with documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases, a blood sample with simultaneous follicle-stimulating hormone > 40 mIU/mL and estradiol < 40 pg/mL [< 147 pmol/L] is confirmatory) are eligible. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods outlined for WOCBP if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of postmenopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their postmenopausal status, they can resume use of HRT during the study without use of a contraception method
* Male patients involved with WOCBP must agree to use a highly effective form of contraception or avoid intercourse from time of screening and throughout the study treatment period and for at least 4 months after the last dose of study treatment. Male patients must not freeze or donate sperm starting at screening and throughout the study period and at least 4 months after the final study treatment administration. Preservation of sperm should be considered prior to enrollment in this study
* Ability to understand and the willingness to sign a written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants
* Willing to undergo biopsy as required by the study (dose expansion only)

Exclusion Criteria:

* As azenosertib (ZN-c3) is a substrate of CYP3A4, use of prescription or non-prescription drugs known to be moderate or strong inhibitors or inducers of CYP3A4 are prohibited with the exception of moderate or strong inhibitors or inducers of CYP3A4 that are part of the prophylactic antiemetic regimen. Chloroquine/hydroxychloroquine are metabolized by CYP3A4 and therefore, should be prohibited. For patients who have received prior moderate or strong inhibitors or inducers of CYP3A4, the required washout period is approximately 5 half-lives prior to study treatment initiation
* Patients who are receiving any other investigational agents
* Patients who have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to the study drugs
* Patients who have a history of severe hypersensitivity reactions to other monoclonal antibodies (mAbs)
* Patients with clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses including, but not limited to, any underlying pulmonary disorder (i.e., pulmonary emboli within 3 months of the study enrollment, severe asthma, severe chronic obstructive pulmonary disease, restrictive lung disease, pleural effusion, etc.), and any autoimmune, connective tissue or inflammatory disorders with potential pulmonary involvement (i.e., rheumatoid arthritis, Sjogren's, sarcoidosis, etc.), or prior pneumonectomy
* Pregnant women are excluded from this study because T-DXd (DS-8201a) and azenosertib (ZN-c3) have the potential risk for teratogenic or abortifacient effects. Because there is an unknown but potential risk for AEs in nursing infants secondary to treatment of the mother with T-DXd (DS-8201a) and azenosertib (ZN-c3), breastfeeding should be discontinued if the mother is treated with T-DXd (DS-8201a) or azenosertib (ZN-c3)
* Patients with history of non-infectious pneumonitis/interstitial lung disease (ILD), current ILD, or where suspected ILD cannot be ruled out by imaging at screening
* Patients with active infections requiring antibiotics at the time of study treatment initiation are not eligible
* Patients with history of malabsorption syndrome or other condition that would interfere with enteral absorption or results in the inability or unwillingness to swallow pills
* Patients with current signs or symptoms of bowel obstruction including sub-occlusive disease related to underlying disease
* Patients with a medical history of myocardial infarction within 6 months before enrollment, symptomatic congestive heart failure (New York Heart Association class IIb to IV), and/or troponin levels consistent with myocardial infarction as defined according to the manufacturer 28 days prior to enrollment
* Patients with clinically significant corneal disease
* Patients with a pleural effusion, ascites, or pericardial effusion that requires drainage, peritoneal shunt, or cell-free and concentrated ascites reinfusion therapy (CART). (Drainage and CART are not allowed within 2 weeks prior to screening assessment)
* Patients with history of Torsades de Pointes unless all risk factors that contributed to Torsades de Pointes have been corrected
* Based on an average of triplicate 12-lead electrocardiogram (ECG), patients with a mean resting corrected QT (QTc) interval using Fridericia formula of > 470 msec for both males and females at screening or a history of congenital long QT syndrome will be excluded
* Patients with prior treatment with a WEE1 inhibitor (dose escalation and dose expansion)
* Patients with prior treatment with T-DXd (DS-8201a) or other topoisomerase inhibitors (dose escalation and dose expansion)
* Patients with uncontrolled intercurrent illness
* Patients with prior allogeneic organ transplantation including allogeneic stem cell transplantation
* Patients with clinically significant chronic gastrointestinal disorder with diarrhea as a major symptom; ≥ grade 2 diarrhea at baseline. Please contact the protocol principal investigator (PI) for any patient with more than two episodes of diarrhea per day averaged over at least a 7-day period at time of screening to determine whether the diarrhea would be considered clinically significant
* Patients with spinal cord compression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2027-07-08 (Estimated); Study Completion 2027-07-08 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose | Up to completion of dose-escalation
  A Bayesian optimal interval design will be used to determine the maximum tolerated dose of the T-DXd (DS-8201a) and azenosertib (ZN-c3) combination.
Recommended phase 2 dose | Up to completion of dose-escalation
Incidence of dose limiting toxicities (DLTs) | Up to completion of dose-escalation
  DLTs will be defined as the below based on the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0.
Incidence of adverse events (AEs) | Up to 30 days after the last administration of study intervention
  The incidence of AEs of the T-DXd (DS-8201a) and azenosertib (ZN-c3) combination, including but not limited to treatment-emergent adverse events, serious adverse events, deaths, and clinical laboratory abnormalities, will be assessed by the NCI CTCAE version 5.0. AEs will be tabulated by grade and by relationship to the study drugs. The proportion of patients who discontinue study treatment due to AEs and the unacceptable toxicity rate will be estimated with a 95% confidence intervals (CIs).

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 3 years
  ORR will be the percentage of patients with complete response (CR) or partial response (PR), as assessed by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. ORR will be estimated with a 95% CIs.
Progression free survival (PFS) | From study treatment initiation to the date of disease progression, assessed up to 3 years
  Disease progression will be assessed by RECIST version 1.1. PFS will be estimated using the product-limit estimator of Kaplan-Meier.
Duration of response | From initial response (CR or PR) to the first date of documented disease progression or death, assessed up to 3 years
  Duration of response will be estimated using the product-limit estimator of Kaplan-Meier.
Pharmacodynamic effects in the tumor | Up to 3 years
  Two-sample t-test (or Wilcoxon rank sum test) or Chi-square test will be used to compare pharmacodynamic markers between the two expansion cohorts.
Predictors of response and acquired resistance | Up to 3 years
  Predictors of response and acquired resistance may include baseline HER2 expression and copy number, cycle E amplification and expression and other genomic co-alterations, and transcriptional and proteomic profile. Logistic regression and Cox proportional hazards model will be used to assess the relationship between clinical responses and molecular and genomic biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Funda Meric-Bernstam, Principal Investigator — University of Texas MD Anderson Cancer Center LAO
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
"NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page."
URL: https://grants.nih.gov/policy/sharing.htm